CLINICAL TRIAL: NCT06564363
Title: The Efficacy of the IUrisure for Detection of Recurrent Urothelial Carcinoma: a Single Center Prospective Study
Brief Title: The Efficacy of the IUrisure for Detection of Recurrent Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan Ammunition Life-tech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BDY003
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-11

CONDITIONS: Urothelial Carcinoma
Keywords: Bladder cancer; Upper tract urothelial carcinomas; Recurrence; Methylation
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urothelial carcinoma Patients: Patients with urothelial carcinoma, which can be primary or recurrent, should be eligible for surgery including transurethral resection of bladder tumours (TURbt), partial cystectomy, radical nephroureterectomy, and kidney-sparing surgery. Urine samples were collected before and after surgery. The follow-up period was 24 months, and the patients underwent routine tests during the follow-up period. The gold standard for recurrence of urothelial carcinoma is surgical/biopsy pathology.
  Interventions: Diagnostic Test: IUrisure test

INTERVENTIONS:
Diagnostic Test: IUrisure test — Postoperative patients are followed up every three months on average, and IUrisure test was performed at each follow-up visit.

SUMMARY:
The clinical trial was designed to determine the efficacy (sensitivity and specificity) of the IUrisure test compared to the gold standard cystoscopy and pathology in patients under monitoring for recurrence of urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high suspicion/confirmed urothelial carcinoma by CT, CTU, MR and other imaging examinations and meet the indications for surgery, including TURbt, partial cystectomy, radical nephroperectomy and kidney-sparing surgery;
2. Patients with highly suspected/confirmed recurrence of urothelial carcinoma who meet the indications for surgery, including TURbt, partial cystectomy, radical nephroperectomy and kidney-sparing surgery;
3. The patient agrees to participate in this study and has signed the informed consent form.

Exclusion Criteria:

* (1) Patients with urothelial carcinoma combined with other malignant tumors; (2) Patients with a history of other non-urothelial carcinoma cancers; (3) Samples that are not urothelial carcinoma in surgical pathology; (4) Samples of Ta/low-grade urothelial carcinoma shown by surgical pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All urothelial carcinoma patients were not Ta stage or low-grade who met the indications for surgery. Surgical modalities include transurethral resection of bladder tumours (TURbt), partial cystectomy, radical nephroureterectomy, and kidney-sparing surgery. Urine samples were collected before and after surgery, and IUrisure methylation test was performed on each urine sample. The follow-up period was 24 months, and the patients underwent routine tests during the follow-up period. The gold standard for recurrence of urothelial carcinoma is surgical/biopsy pathology.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Specificity of IUrisure test | Day 1
  The proportion of negatives that are correctly identified as such by the gold standard
Sensitivity of IUrisure test | Day 1
  The proportion of positives that are correctly identified as such by the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China